CLINICAL TRIAL: NCT05799586
Title: Traditional Chinese Medicine Health Preservation Intervention for Depression: A Pilot Randomized Controlled Trial
Brief Title: TCM Health Preservation for Depression
Acronym: TCMHPFD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TCMHPFD; No.21B2/004A (Other Grant/Funding Number: the Chinese Medicine Development Fund, Hong Kong Special Administrative Region, China)
Record Dates: First submitted 2023-03-23; First posted 2023-04-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-03

CONDITIONS: Depressive, Symptoms Depressive Disorder, Depression
Keywords: Depression; Traditional Chinese Medicine; Randomized Controlled Trial; Health preservation
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Two-arm parallel assignment involves two groups of participants. In this study, one group will receive Traditional Chinese Medicine health preservation for depression, and the other group will receive the waitlist control. Thus, during the trial, participants in one group receive Traditional Chinese Medicine health preservation "in parallel" to participants in the waitlist control group.
Who Masked: Outcomes Assessor
Masking Description: The researchers who perform the outcome measurement and those researchers who conduct data analysis will be blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional Chinese medicine health preservation group (Experimental): The participants in the traditional Chinese medicine health preservation group will attend six traditional Chinese medicine health preservation courses (2h each per one, for 6 weeks) to learn and experience traditional Chinese medicine health preservation from a registered traditional Chinese medicine practitioner in a classroom at the School Nursing, the Hong Kong Polytechnic University.
  Each class will be conducted in a small group of 4 to 6 participants to enhance interaction and ensure the quality of teaching. Participants will then practice traditional Chinese medicine health preservation at home for 6 weeks.
  Interventions: Behavioral: Traditional Chinese Medicine health preservation group; Behavioral: Waitlist control group
- Waitlist control group (No Intervention): Participants in the waitlist control group will receive usual care during the 6-week waitlist period of intervention, and 6-week waitlist period of follow-up. After the follow-up assessment, they will be provided an equivalent traditional Chinese medicine health preservation for depression.

INTERVENTIONS:
Behavioral: Traditional Chinese Medicine health preservation group — The traditional Chinese medicine health preservation intervention for depression was developed based on a previous systematic review and meta-analysis of Traditional Chinese medicine based integrated health interventions for depression, traditional Chinese medicine health preservation textbooks, clinical practice guidelines related to traditional Chinese medicine health preservation and traditional Chinese medicine treatment for depression. The content and structure of traditional Chinese medicine health preservation for depression was achieved among Hong Kong traditional Chinese medicine experts via a Delphi study.
  Arms: traditional Chinese medicine health preservation group
Behavioral: Waitlist control group — Usual care
  Arms: traditional Chinese medicine health preservation group

SUMMARY:
This study aims to evaluate the feasibility and preliminary effects of Traditional Chinese Medicine (TCM) health preservation for depression on depressive symptoms reduction and other health-related outcomes among Hong Kong Chinese adults with depression. Participants in intervention group will receive TCM health preservation course for six weeks (6 sessions, 2 hours each) and practice TCM health preservation during the 6-week follow-up period. Participants in the control group (waitlist control) will receive usual care. After the follow-up assessment, TCM health preservation courses for depression will be provided to them for compensation.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong Chinese adults aged 18-years-old to 65-years-old;
* diagnosed with moderate level of depression (a score of 10~20), evaluated by the Patient Health Questionnaire-9 (PHQ-9);
* can communicate in spoken Cantonese and written Chinese;
* willing to provide written informed consent and be able to adhere to the study protocol.

Exclusion Criteria:

* being pregnant or during the lactation, or plan to get pregnant;
* new onset or change of antidepressant medication or dosage in the last 3 months;
* PHQ-9 score≥20, meaning a severe level of depression;
* with a previous or present diagnosis of psychotic disorders as screened by the Chinese version of the Structured Clinical Interview for DSM-IV;
* the score of Hong Kong Montreal Cognitive Assessment less than 22;
* significant suicidal risk as rated by the Hamilton Depression Rating Scale item on suicide (score ≥3);
* with diagnosis of illness which can interfere the individuals to participate or adhere to the modified lifestyle;
* with diagnosis of medical conditions, which are not suitable to modify diet or do physical activities recommended by physicians;
* joining in another clinical trial during the study period;
* with any major medical condition that causes depression based on the judgement of the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Change in the Patient Health Questionnaire (PHQ-9) | Time Frame: Baseline, week 2, week 4, week 6, week 8, week 12
  The PHQ-9, a self-rated questionnaire to assess the presence and severity of depressive symptoms of an individual during the last 2 weeks on a scale of 0 (not at all) to 3 (nearly every day), with a total score ranging from 0 to 27. A higher score indicates a higher severity of depression symptoms.

SECONDARY OUTCOMES:
Change in the Generalized Anxiety Disorder-7 (GAD-7) | Time Frame: Baseline, week 2, week 4, week 6, week 8, week 12
  The GAD-7 is a four-point Likert scale for identifying probable cases of GAD and assess the severity of symptoms of GAD for the past 2 weeks. The total score of GAD-7 varies from 0 to 21, and responses include "nearly every day," "more than half the days," "several days", and "not at all". The cutoff point of 5, 10, and 15 of GAD-7 might be interpreted as showing mild, moderate, and severe levels of anxiety. Higher scores indicate more severe GAD symptoms.
Change in the Perceived Stress Scale (PSS-10) | Time Frame: Baseline, week 2, week 4, week 6, week 8, week 12
  The PSS-10 is a 10-item scale that is often used for measuring perceived psychological stress. Each item is rated on a 5-point Liket scale during the past month, referring to "4" as "very often" and "0" as never. The total score changes from 0 to 40, with a higher score meaning a higher perceived psychological stress level.
Change in the Insomnia Severity Index (ISI) | Time Frame: Baseline, week 2, week 4, week 6, week 8, week 12
  The ISI is a seven-item self-rating scale to assess the severity of insomnia, distress, and functional impairment associated with insomnia on a 5-point Likert scale. The score of each item of ISI ranges from 0 (no problem) to 4 (very severe problem), and the total score is interpreted as below: absence of insomnia as 0 to 7, sub-threshold insomnia as 8 to14, moderate insomnia as 15 to 21, and severe insomnia as 22 to 28.
Change in the Fatigue Assessment Scale (FAS) | Time Frame: Baseline, week 2, week 4, week 6, week 8, week 12
  The FAS is a 10-item scale that evaluates symptoms of chronic fatigue with a five-point Likert-type scale, which ranges from 1 ("never") to 5 ("always"). A higher score means greater fatigue severity. The total score ranges from 10 to 50. A total FAS score < 22 means no fatigue, a score≥ 22 refers to fatigue.
Change in the Short-Form (six-dimension) Health Survey (SF-6D) | Time Frame: Baseline, week 6, week 8, week 12
  The SF-6D covers six domains using a scale of 1 to 6 to evaluate participants' general health and quality of life. Higher scores indicate better health status.
Change in the General Self-Efficacy Scale (GSE) | Time Frame: Baseline, week 2, week 4, week 6, week 8, week 12
  The GSE scale is a four-point Likert scale with ten items appropriate for evaluating an individual's self-efficacy. It is scored ranging from 1 point to 4 points, referring to "not at all true" to "exactly true" and the total score varied from 10 to 40. A higher score shows a more satisfactory self-efficacy.
Change in the Health-Promoting Lifestyle Profile II (HPLP II) | Time Frame: Baseline, week 4, week 6, week 8, week 12
  The HPLP II is a scale with 52 items and 6 domains for measuring health-promoting behavior, defined as a multidimensional pattern of self-initiated perceptions and actions that serve to maintain or increase the level of self-actualization, wellness, and fulfillment of a person. The total scores of HPLP-II varies from 52 to 208. Higher HPLP II score denotes better level of health-promoting lifestyle.

OTHER OUTCOMES:
Change in the Credibility/ Expectancy Questionnaire (CEQ) | Time Frame: Baseline, week 6
  The CEQ is a self-reported scale with 6 items and two subscales of treatment credibility and outcome expectancy to measure the participants' treatment credibility and outcome expectancy for improvement. The final scoring of the CEQ is computed by the sum of the items composing each subscale, with a higher quotation referring to higher treatment credibility and outcome expectation.
  The CEQ taps on participants' affective and cognitive evaluations of treatment satisfaction, credibility, and expectation. The subscale of credibility assesses beliefs about the treatment strength. The expectancy subscale assesses how participants perceive their symptoms will improve during the intervention period.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Nursing, the Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data will be available when the study has been published. The individual participant data will be available upon request.
Supporting Information: Study Protocol, SAP
Time Frame: No time restriction for the data availability
Access Criteria: The individual participant data will be available upon request

REFERENCES:
- [Derived] Ruan JY, Chen X, Cheng HL, Qing WY, Ho JYS, Chen HY, Luo D, Hu L, Chen JY, Wu LY, Chak KY, Lu C, Mak YW, Yeung WF. Perceptions and experiences of a multicomponent traditional Chinese medicine lifestyle medicine program for depression: a qualitative study. BMC Complement Med Ther. 2026 Jan 15. doi: 10.1186/s12906-025-05217-x. Online ahead of print. PMID 41540402